CLINICAL TRIAL: NCT00516646
Title: A Double-blind, Placebo-controlled, Randomized Trial Evaluating the Efficacy and Safety of Alagebrium (ALT-711) in Patients With Chronic Heart Failure
Brief Title: The BENEFICIAL Study: Evaluating the Efficacy and Safety of Alagebrium (ALT-711) in Patients With Chronic Heart Failure
Acronym: BENEFICIAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synvista Therapeutics, Inc (Industry)
Responsible Party: A.A. Voors, MD PhD, University Medical Center Groningen, Groningen, The Netherlands
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALT-711-0527
Record Dates: First submitted 2007-08-13; First posted 2007-08-15 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-04

CONDITIONS: Heart Failure
Keywords: Advanced Glycation End-products (AGEs); Alegebrium
MeSH Terms: conditions — Heart Failure | interventions — alagebrium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): ALT-711 200 mg bid
  Interventions: Drug: ALT-711
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALT-711 — 200 mg bid
  Other Names: Alagebrium
  Arms: 1
Drug: Placebo — bid
  Arms: 2

SUMMARY:
Several lines of evidence have suggested that Advanced Glycation End-products (AGEs) play a role in the development and progression of heart failure. The AGE-crosslink breaker Alagebrium (ALT-711) improved cardiac function and symptoms in experimental and small human heart failure studies. These results have not yet been confirmed in a randomized controlled clinical trial.

DETAILED DESCRIPTION:
This study is a double-blind, randomized, placebo-controlled, parallel design trial enrolling 100 patients (2x50) with stable CHF. Patients will be randomized to either 200 mg Alagebrium twice daily or placebo for a period of 9 months. Efficacy measurements will be performed at baseline, and at the end of the study, and include aerobic capacity (VO2max) exercise testing, echocardiography, Minnesota Living with Heart Failure score, AGEs measurements in blood and skin, NYHA heart failure class, patient's and physician's global assessment, and levels of NT-pro-BNP. Safety visits are performed at 3 months intervals. In addition, one safety visit will be performed 2 weeks after the randomization visit and 1 month after the last treatment visit. A total of 8 visits will be performed during the entire study.

ELIGIBILITY:
Inclusion Criteria:

* NYHA II-IV heart failure
* Echocardiographic ejection fraction ≤ 40%
* Duration of heart failure > 3 months
* Stable heart failure medical therapy for > 1 months

Exclusion Criteria:

* History of myocardial infarction in previous 6 months
* History of stroke in previous 6 months
* Clinically significant renal, liver, pulmonary,or hematological disease
* Active and or treated malignancies within 12 months
* Uncontrolled diabetes mellitus

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary end-point of the study will be aerobic capacity (VO2max) measured at exercise testing | At baseline and after 9 months of study drug

SECONDARY OUTCOMES:
Changes in systolic function, diastolic function, advanced glycation end-products (AGE) measurements, changes in Minnesota Living with Heart Failure score, NYHA heart failure score, patient's and physician's global assessment, and NT-pro-BNP | At baseline and after 9 months of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan A Voors, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (1):
- Dept. Cardiology - University Medical Center Groningen, Groningen, P.O. Box 30 001, Netherlands

REFERENCES:
- [Background] Thohan V, Koerner MM, Pratt CM, Torre GA. Improvements in Diastolic Function Among Patients with Advanced Systolic Heart Failure Utilizing Alagebrium (an Oral Advanced Glycation End-product Cross-link Breaker). American Heart Association Scientific Sessions . 2005. Ref Type: Abstract
- [Background] Little WC, Zile MR, Kitzman DW, Hundley WG, O'Brien TX, Degroof RC. The effect of alagebrium chloride (ALT-711), a novel glucose cross-link breaker, in the treatment of elderly patients with diastolic heart failure. J Card Fail. 2005 Apr;11(3):191-5. doi: 10.1016/j.cardfail.2004.09.010. PMID 15812746
- [Derived] Hartog JW, Willemsen S, van Veldhuisen DJ, Posma JL, van Wijk LM, Hummel YM, Hillege HL, Voors AA; BENEFICIAL investigators. Effects of alagebrium, an advanced glycation endproduct breaker, on exercise tolerance and cardiac function in patients with chronic heart failure. Eur J Heart Fail. 2011 Aug;13(8):899-908. doi: 10.1093/eurjhf/hfr067. Epub 2011 Jun 13. PMID 21669961
- [Derived] Willemsen S, Hartog JW, Hummel YM, Posma JL, van Wijk LM, van Veldhuisen DJ, Voors AA. Effects of alagebrium, an advanced glycation end-product breaker, in patients with chronic heart failure: study design and baseline characteristics of the BENEFICIAL trial. Eur J Heart Fail. 2010 Mar;12(3):294-300. doi: 10.1093/eurjhf/hfp207. Epub 2010 Jan 25. PMID 20100811